CLINICAL TRIAL: NCT00994721
Title: A Randomized Phase III Study of Adjuvant Gemcitabine Versus Gemcitabine Plus Concurrent Chemoradiation in Pancreatic Cancer Underwent Curative Intent (R0 / R1) Resection
Brief Title: A Phase III Study of Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Chang Gung Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Mackay Memorial Hospital (Other); Taichung Veterans General Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Veterans General Hospital. (Other); Kaohsiung Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: T3207
Record Dates: First submitted 2008-03-26; First posted 2009-10-14 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2009-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pancreatic cancer: resected pancreatic cancer

SUMMARY:
Study Design： Adjuvant gemcitabine therapy has been shown to improve recurrence-free survival in pancreatic cancer underwent curative intent resection. This study is to evaluate whether combining concurrent chemo-radiotherapy can further improve the recurrence-free survival benefit of adjuvant gemcitabine chemotherapy in pancreatic cancer underwent curative resection.

Research Objective and Study End Points

1. Primary endpoint： The primary end point is disease free survival.
2. Secondary endpoints： The secondary end points are to evaluate the overall survival, local and distant recurrence rate, and impact on quality of life after adjuvant gemcitabine with or without CCRT in curatively resected pancreatic cancer.

Furthermore, the clinical, pathological and molecular prognostic factors in curatively resected pancreatic cancers will be evaluated.

DETAILED DESCRIPTION:
Treatment plan and Randomization scheme:：

Patients will be randomized after stratification according to pathology report on section margin, tumor size, lymph node metastasis:

Patients who are randomized to Arm 1 will receive adjuvant chemotherapy started within 4-8 weeks after the surgery, and administered at D1, D8 and D15 every 4 weeks for 6 cycles (6 months). Patients who are allocated to Arm 2 will receive sandwich treatment, which comprised of the same adjuvant chemotherapy within 4-8 weeks after the surgery for 3 cycles (3 months), followed by CCRT (start 4-6 weeks after the last dose of 3rd cycle chemotherapy) and then another 3 cycles of gemcitabine monotherapy.

Statistical Consideration:

We anticipate the 2-year disease free survival will increase from 25% to 40% with the incorporation of CCRT into the adjuvant treatment for post-operative pancreatic adenocarcinoma. With a significant level of 0.05, 107 patients will be required for each treatment arm to reach 80% statistical power. Since the drop out rate is approximately 10%, 265 patients will be enrolled to ensure that we will have 214 (107x2) eligible patients in this study. We anticipate that we will recruit roughly 67 patients per year, therefore, patient recruitment will be completed in 4 years.

Randomization scheme:

Histo-/cyto-logically confirmed macroscopic complete resected pancreatic adenocarcinoma

1. The primary end-point is disease free survival.
2. The secondary end-points are overall survival; local and distant control rate, and the quality of life.
3. The clinical and molecular prognostic factors for overall survival.

   * Radiation fields encompass initial main tumor of pancreas only with a safe margin of 1cm. Lymph node regions initially involved with tumor confirmed by excision will be included in the clinical target volume. Elective radiation to uninvolved lymph nodes will not be given.

ELIGIBILITY:
A.Eligibility Criteria

1. Patients with pancreatic cancer after curative intent resection.
2. The histology of resected tumor has to be adenocarcinoma.
3. Age 20-75 years.
4. ECOG performance scale 0-1.
5. Patients must have normal organ and marrow function as defined below.
6. The effects of study agents on the developing human fetus at the recommended therapeutic dose are unknown.
7. to sign a written informed consent.
8. Registered within 6 weeks after surgery.
9. Preoperative abdominal CT or MRI with contrast enhancement.

B.Exclusion Criteria

1. Patients with gross residual, macroscopic positive resection margin or distant metastases.
2. Patients may not be receiving any other investigational agents.
3. Patients who have had prior chemotherapy or radiotherapy are not eligible.
4. History of allergic reactions.
5. Patients who had non-curable second primary malignancy.
6. Uncontrolled intercurrent illness including.
7. Pregnant women.
8. receiving immuno-suppressive therapy、anti-coagulants.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We anticipate the 2-year disease free survival will increase from 25% to 40% with the incorporation of CCRT into the adjuvant treatment for post-operative pancreatic andenocarcinoma. With a significant level of 0.05,107 patients will be required for each treatment arm to reach 80% statistical power. Since the drop out rate is approximately 10%, 265 patients will be enrolled to ensure that we will have 214(107x2) eligible patients in this study. We anticipate that we will recruit roughly 67 patients per year, therefore, patient recruitment will be completed in 4 years.
Sampling Method: Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2009-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The primary end-point is recurrence-free survival. | Pancreatic Cancer Disease Committee

SECONDARY OUTCOMES:
The secondary end-points are overall survival; local and distant control rate, and the quality of life. | Pancreatic Cancer Disease Committee

CONTACTS AND LOCATIONS:
Overall Officials: Tsann-Long Hwang, M.D., Study Chair — Chang Gung Memorial Hospital; Yu-Wen Tien Tien, Ph.D., Principal Investigator — National Taiwan University Hospital; Yi-Ming Shyr, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan; Pin-Wen Lin, M.D, Principal Investigator — National Cheng-Kung University Hospital; Yu-Lin Lin, M.D., Principal Investigator — National Taiwan University Hospital
Locations (3):
- Taiwan (3):
  - Chang-Gung Memorial Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiu YF, Liu TW, Shan YS, Chen JS, Li CP, Ho CL, Hsieh RK, Hwang TL, Chen LT, Ch'ang HJ; Taiwan Cooperative Oncology Group pancreatic cancer study group. Carbohydrate Antigen 19-9 Response to Initial Adjuvant Chemotherapy Predicts Survival and Failure Pattern of Resected Pancreatic Adenocarcinoma but Not Which Patients Are Suited for Additional Adjuvant Chemoradiation Therapy: From a Prospective Randomized Study. Int J Radiat Oncol Biol Phys. 2023 Sep 1;117(1):74-86. doi: 10.1016/j.ijrobp.2023.02.061. Epub 2023 Apr 11. PMID 37055279